CLINICAL TRIAL: NCT01819831
Title: A Phase II Trial of Preoperative Proton Therapy in Soft-tissue Sarcomas of the Extremities and Body Wall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gary Yang, MD, Principal Investigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5120263
Record Dates: First submitted 2013-03-18; First posted 2013-03-28 (Estimated); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: extremity soft tissue sarcoma; proton radiation; preoperative radiation
MeSH Terms: conditions — Sarcoma | interventions — Proton Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Preoperative proton radiation (Experimental): Patients will receive 50 Gray equivalents (GyE) in 25 fractions with proton therapy, followed by surgery 4-8 weeks after completion of radiation.
  Interventions: Radiation: proton radiation; Procedure: surgery (wide local excision; limb preservation surgery)

INTERVENTIONS:
Radiation: proton radiation — proton radiation: 2 GyE/Day to isocenter, one treatment per day, 5 days per week for 25 treatments (=50 GyE to isocenter/25 fractions)
  Other Names: Proton radiotherapy; Proton treatment
Procedure: surgery (wide local excision; limb preservation surgery) — In areas with ample soft tissue that can be removed without compromising future function or wound closure, wide margins is the goal of treatment; associated rates of local failure are low in such instances. Margins will be determined by the surgeon; the goal is to achieve at least a 2 mm negative margin resection. However, smaller margins can be acceptable if it allows for limb-sparing surgery with conserved functional outcomes. Every effort will be made to have limb preservation surgery unless there is documented evidence of tumor progression during or after the course of radiation that would require amputation for an appropriate margin resection.
  Other Names: wide local excision; limb preservation surgery

SUMMARY:
When treated with surgery alone, many soft-tissue sarcomas have a high chance of coming back. Radiation therapy is frequently used in addition to surgery to reduce the chances of the sarcoma coming back. However, radiation can have long-term side effects on the normal tissues surrounding the tumor, leading to problems such as swelling, scarring, and joint stiffness.

Recently, there have been advances in the way that radiation therapy can be given. Proton radiation therapy is one of those advances. With proton radiation, it is possible to give radiation over a smaller area surrounding the tumor, resulting in less radiation to the surrounding normal tissues.

The purpose of this study is to determine whether proton radiation decreases the long-term side effects of radiation on normal tissues and if smaller proton radiation fields reduce local recurrence compared to the larger radiation fields that have been used in prior studies.

DETAILED DESCRIPTION:
Data support preoperative radiotherapy as one of the standard options in the management of large or high-grade extremity soft tissue sarcomas (STS). The advantages of preoperative radiotherapy are lower doses and smaller radiation volumes; these may be used to effect improvement of long-term side effects and extremity function. Another potential advantage is assisting surgery through tumor shrinkage and reduction of tumor cell seeding. The disadvantage of preoperative radiation is the higher likelihood of postoperative wound complications, but in a prospective phase III trial these complications were found to be generally temporary and without significant effect on long term function.

Combined conservative surgery and radiotherapy has shown to achieve excellent local control in sarcoma patients following margin-negative surgery, but late radiation morbidity and reduced quality of life may result from adjuvant radiation. The dosimetric advantage of proton radiotherapy may translate into reduced acute and late effects due to improved normal-tissue sparing in the treatment of extremity and truncal STS. However, these potential advantages need to be validated in clinical trials. The investigators propose a phase II study to evaluate the effect of preoperative proton radiotherapy on the reduction of late radiation morbidity, patterns of failure, and impact of late radiation morbidity on general quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary soft tissue sarcoma of the upper extremity (including shoulder), lower extremity (including hip) or body trunk (excluding retroperitoneum).
* No clinical evidence of distant metastatic disease
* Evaluation by surgeon, with documentation that the tumor is resectable
* ECOG performance status 0-1
* For females of childbearing potential, a serum pregnancy test within 4 weeks prior to registration
* Patient must practice adequate contraception
* Adequate bone marrow function

Exclusion Criteria:

* Patients with sarcoma of the head, neck, intra-abdominal or retroperitoneal region, hand or foot
* Histopathology demonstrating rhabdomyosarcoma, extraosseous primitive neuroectodermal tumor (PNET), soft tissue Ewing's sarcoma, osteosarcoma, Kaposi's sarcoma, angiosarcoma, aggressive fibromatosis, dermatofibrosarcoma protuberans or chondrosarcoma
* Clinical evidence of regional lymph node or distant metastatic disease
* Prior invasive malignancy (except non-melanomatous skin cancer or early stage prostate cancer) unless disease free for a minimum of 3 years
* Prior radiotherapy to the potential target anatomic region would result in overlap of radiation fields for current sarcoma
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to used medically acceptable forms of contraception

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Yang, MD, Principal Investigator — gyang@llu.edu
Locations (1):
- Loma Linda University Medical Center / James M. Slater Proton Treatment Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Proton Radiation
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Late Radiation Toxicities at 2 Years From the Start of Radiation Treatment
Description: To report the number of participants with late radiation morbidity
  Late subcutaneous fibrosis and joint stiffness are assessed using the European Organization for Research and Treatment of Cancer/Radiation Therapy Oncology Group (EORTC/RTOG) late toxicity scoring criteria below:
  Subcutaneous tissue: Grade 1(slight fibrosis; subcutaneous fat loss), Grade 2(moderate fibrosis: slight field contracture), Grade 3(severe fibrosis; field contracture >10%), Grade 4(necrosis), Grade 0 (none) Joint stiffness: Grade 1(mild stiffness; slight range of motion loss), Grade 2(Moderate stiffness, pain, range of motion loss), Grade 3(Severe stiffness, pain, range of motion loss), Grade 4(necrosis; complete fixation), Grade 0 (none) Lymphedema is measured according to the criteria of Stern: Score 0(none), Score 1(Mild but definite swelling), Score 2(Moderate), Score 3(Severe, considerable swelling), Grade 4(Very severe (skin shiny & tight)
Time Frame: at 2 years from the start of radiation treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Grade 3-5 Adverse Events at 6 Months From the Start of Radiation Treatment.
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for reporting of adverse events.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Patterns of Failure at 6 Months From the Start of Radiation Treatment
Description: Prespecified patterns of failure, including local failure, regional failure, distant failure, and death without disease progression at 6 months from the start of radiation treatment measured by CT or MRI scan
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Patterns of Failure at 6 Months
Description: Patterns of failure including local failure, distant failure, distant-disease-free survival, disease-free survival, overall survival rates, and second primary tumor at 6 month from the start of radiation treatment on CT or MRI scan.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
participants
  local failure | 0
  distant failure | 1
  distant-disease-free survival | 5
  disease-free survival | 5
  overall survival | 6
  second primary tumor | 0

5. Secondary Outcome: Wound Complication Rates Infection, Dehiscence at 6 Months From the Start of Radiation Treatment.
Description: Wound complications - Major wound complications, such as secondary operations, re-admissions, and/or invasive procedures for wound complication (deep wound packing and/or prolonged dressing changes) due to Infection, dehiscence.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 6
Participants | 1

6. Secondary Outcome: Report of Late Radiation Morbidity at 2 Years
Description: To report the number of participants with late radiation morbidity using quality of life survey including physical, emotional, social/family and functional well-being.
Time Frame: at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Proton Radiation
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: At 6 months and 2 years post-enrollment.
Arm/Group | Preoperative Proton Radiation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative Proton Radiation (N=6)
dehiscence (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT01819831/Prot_SAP_000.pdf